CLINICAL TRIAL: NCT01827072
Title: NPB-01(Intravenous Immunoglobulin) Maintenance Therapy for Patients With Multifocal Motor Neuropathy.
Brief Title: Phase III Clinical Trial of NPB-01maintenance Therapy in Patients With Multifocal Motor Neuropathy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nihon Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPB-01-10/C-01
Record Dates: First submitted 2013-04-01; First posted 2013-04-09 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2014-10

CONDITIONS: Multifocal Motor Neuropathy
Keywords: IVIG in Multifocal Motor Neuropathy; Patients with Multifocal Motor Neuropathy
MeSH Terms: interventions — Immunoglobulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NPB-01 (Experimental): Intravenous immunoglobulin
  Interventions: Drug: NPB-01

INTERVENTIONS:
Drug: NPB-01
  Other Names: immunoglobulin

SUMMARY:
Patients diagnosed with Multifocal Motor Neuropathy were confirmed based on the European Federation of Neurological Societies/ Peripheral. Nerve Society Guideline. Patients who meet all inclusion criteria and do not conflict with the exclusion criteria will receive NPB-01 (intravenous immunoglobulin) 400mg/kg/day for five consecutive days. Subsequently, patients receive NPB-01 1g/kg every 3weeks and evaluate the Medical Research Council（MRC） score and the Guy's Neurological Disability Scale（GNDS） et al.

As a safety endpoint, the safety of NPB-01 will be investigated the occurrence of adverse events by one year after the start of the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who need high-dose intravenous immunoglobulin（greater than or equal to 1g/kg） therapy.
* 2. Patients who continued treatment for MMN without addition or increase at 30 days before informed consent.
* 3. Patients who MRC score increased 1 stage in greater than or equal to 2 muscles and not decreased relative other muscles to before at after in high-dose intravenous immunoglobulin therapy.
* 4. Patients with greater than or equal to twenty years old at informed consent.

Exclusion Criteria:

* 1. Patients treated with Plasmapheresis at 3 months before informed consent.
* 2. Patients treated with Rituximab or Natalizumab at 6 months before informed consent.
* 3. Patients treated with Interferon-beta at 6 months before informed consent.
* 4. Patients treated with high-dose intravenous immunoglobulin（greater than or equal to 1g/kg） at 8 weeks before informed consent.
* 5. Patients treated with intravenous immunoglobulin at 3 weeks before informed consent.
* 6. Patients with history of shock or hypersensitivity for NPB-01.
* 7. Patients with IgA deficiency.
* 8. Patients with malignancy.
* 9. Patients with impaired liver function.
* 10. Patients with impaired renal function.
* 11. Patients with cerebro- or cardiovascular disorders.
* 12. Patients with high risk of thromboembolism.
* 13. Patients with hemolytic/hemorrhagic anemia.
* 14. Patients with decreased cardiac function.
* 15. Patients with decreased platelet.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Medical Research Council（MRC） score | 49 weeks
maximum grip strength | 49 weeks
The Guy's Neurological Disability Scale (GDNS) | 49 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Nihon Pharmaceutical Co., Ltd, Osaka, Japan

REFERENCES:
- [Derived] Kuwabara S, Misawa S, Mori M, Iwai Y, Ochi K, Suzuki H, Nodera H, Tamaoka A, Iijima M, Toda T, Yoshikawa H, Kanda T, Sakamoto K, Kusunoki S, Sobue G, Kaji R; Glovenin-I MMN Study Group. Intravenous immunoglobulin for maintenance treatment of multifocal motor neuropathy: A multi-center, open-label, 52-week phase 3 trial. J Peripher Nerv Syst. 2018 Jun;23(2):115-119. doi: 10.1111/jns.12268. Epub 2018 Apr 24. PMID 29635876